CLINICAL TRIAL: NCT04621955
Title: Observational Study of Home Administration of Carfilzomib: Feasibility, Quality of Life and Description of the Process With Related Health-care Economics
Brief Title: Observational Study of Home Administration of Carfilzomib
Acronym: KARE-2
Status: Withdrawn | Type: Observational
Why Stopped: Not possible to conduct study
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 20167745
Record Dates: First submitted 2017-05-02; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma; Hematologic Diseases
Keywords: Home administration of chemotherapy; Relapsed and/or refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the feasibility of an at home administration program for carfilzomib patients.

DETAILED DESCRIPTION:
In this observational study, the feasibility of an at home administration program for carfilzomib will be evaluated in patients with relapsed and/or refractory multiple myeloma having already received a minimum of 2 and a maximum of 6 full cycles of KRd (carfilzomib - lenalidomide - dexamethasone) in the hospital.

One treatment cycle of KRd consists of a 28-day period. Carfilzomib is administered intravenously as a 10 minute infusion, on two consecutive days, each week for three weeks (days 1, 2, 8, 9, 15 and 16), followed by a 12-day rest period (days 17 - 28). In combination with carfilzomib, lenalidomide is administered orally on days 1-21 and dexamethasone is administered orally on days 1, 8, 15 and 22 of the 28-day cycles.

Multiple myeloma is characterized by a recurring pattern of remission and relapse. Given the need for chronic treatment and good adherence, convenience and quality of life of the patients become important factors as well. As the majority of the multiple myeloma patients are elderly and the treatment schedule requires many hospital visits, this treatment schedule may impact the social and familial life of the patient.

If the patient accepts to participate in the home administration program:

* Administration of carfilzomib during cycle 1 and 2 will be performed in the hospital
* During cycle 3 until 6, carfilzomib will be administered on day 1 and15 in the hospital, while there will be home administration on days 2, 8, 9 and 16.
* On day 1 of each cycle, there will be asked to the patient to complete a short questionnaire about the quality of life and patients satisfaction during the home administration program of carfilzomib.

If the patient doesn't accept to participate in the home administration program:

-The patient can agree on one-time collection of data: patient characteristics (date of birth+gender) and reason for refusal to the home administration program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to understand the informed consent and willingness to provide an informed consent signature
* Signed and dated written informed consent available (for participation in the home administration program or for agreement on data-collection in case of refusal to participate (reasons for refusal))
* Diagnosis of a relapsed and/or refractory multiple myeloma (refractory meaning nonresponsive (stable or progressive disease) during treatment or disease progression within 60 days of treatment discontinuation)
* Patient on KRd treatment (according to reimbursement criteria) having already received a minimum of 2 and a maximum of 6 full cycles of KRd in the hospital
* Patient with good tolerance of KRd and expected to receive ≥ 6 cycles based on clinical assessment of the treating physician
* Patient willing to receive at home intravenous administration of carfilzomib (only for patients who accepted the home administration program of the study)

Exclusion Criteria:

* Lactating or pregnant females
* Women of childbearing potential unless all of the conditions of the Pregnancy Prevention Program of lenalidomide are met and unless use effective contraception measures during and for one month following treatment. Male patients should use contraception and refrain form sperm donation for at least 90 days after the last dose of carfilzomib.
* Patients who already received carfilzomib home administration
* Any contra-indication for continuation of treatment with carfilzomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients on KRd treatment
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Description of feasibility of home administration | through study completion
  Percentage of patients still in the home administration program 4 cycles mixed home/hospital and who did not discontinue due to AE (adverse event) or PD (progressive disease)

SECONDARY OUTCOMES:
Description of quality of life/satisfaction of the program | through study completion
  Quality of life and satisfaction of the program during home administration of carfilzomib evaluation via "a validated QoL questionnaire on day 1 of each cycle"
Description of patients acceptability | At screening
  Evaluation of percentage of patients who have accepted or refused to enter the home infusion program and reasons of refusal if so.
Description of patient characteristics: performance status | through study completion
  Description of performance status (via Karnofsky scaling)
Description of patient characteristics: professionally active at diagnosis | At screening
  Percentage of patients professionally active at time of diagnosis of multiple myeloma
Description of patient characteristics: professionally active at study entry | At screening
  Percentage of patients professionally active at study entry
Description of patient characteristics: change of professional activity during study | Through study completion
  Percentage of patients with change in professional activity during study
Description of patients characteristics: extra medical consultations | through study completion
  Description of extra medical consultations (general practitioner, hospitalisations, REMEDUS) and reasons for these visits
Description of the home administration program: reason for discontinuation | through study completion
  Description of reason of discontinuation of home administration program
Description of the home administration program: number of administrations | through study completion
  Description of number of home administrations received vs planned per patient and total population + reasons of missed doses
Description of the home administration program: patients in home infusion program | through study completion
  Percentage of patients still in the home administration program after 2 cycles in the hospital and 4 cycles combined at hospital/at home (full population), whatever the reason for discontinuation
Description of safety: adverse events and serious adverse events (according to CTCAE 4.0) | through study completion
  Incidence, relationship and severity of adverse events, serious adverse events, adverse events leading to discontinuation and adverse events leading to treatment interruption according to CTCAE v4.03 criteria; safety will be reported at home and in the hospital
Description of the cost of at home administration versus hospital administration | Through study completion
  Description of the cost of at home administration versus hospital administration. The cost will be carried out taking into consideration the laws governing the Belgian health care system, in which 100% of cancer medical costs are funded by the government (no expense is charged to the patient), and included all expenditures.
Description of the questionnaire, completed by the physician, to assess his/her opinion on the feasibility and satisfaction of the home administration program | through study completion
  Description of the survey for the principal investigator (completed before and after the study) to give feedback on the home administration program

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, Principal Investigator — UZ Leuven Gasthuisberg
Locations (5):
- Belgium (5):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège, Liège
  - Clinique Saint-Pierre Ottignies, Ottignies
  - AZ Nikolaas, Sint-Niklaas